CLINICAL TRIAL: NCT01911364
Title: A 52-wk Randomized Double Blind Parallel Trial: Combination of Beclometasone+Formoterol+Glycopyrrolate vs Tiotropium and vs Combination of Beclometasone+Formoterol and Tiotropium in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of Fixed Combination of Beclometasone + Formoterol + Glycopyrrolate in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1208-PR-0090; 2013-000063-91 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Frequent exacerbators
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BDP/FF/GB (Experimental): CHF 5993 pMDI 100/6/12.5 mcg 2 inhalations b.i.d
  Interventions: Drug: BDP/FF/GB
- Tiotropium (Active Comparator): Tiotropium bromide 18 mcg
  Interventions: Drug: Tiotropium
- BDP/FF + Tiotropium (Active Comparator): BDP/FF pMDI 100/6/12.5 mcg 2 inhalations b.i.d and Tiotropium 18 mcg daily
  BDP/FF/GB versus BDP/FF + Tiotropium
  Interventions: Drug: BDP/FF + Tiotropium

INTERVENTIONS:
Drug: BDP/FF/GB — Superiority over Tiotropium
  Other Names: CHF 5993 pMDI 100/6/12.5 mcg
  Arms: BDP/FF/GB
Drug: Tiotropium — Superiority of CHF5993 over Tiotropium
  Other Names: Spiriva 18 mcg 1 capsule o.d
  Arms: Tiotropium
Drug: BDP/FF + Tiotropium — non inferiority vs CHF5993
  Other Names: Foster 100/6 mcg 2 inhalations bid + Spiriva 18 mcg o.d.
  Arms: BDP/FF + Tiotropium

SUMMARY:
The purpose of this study is to determine the triple combination of beclometasone dipropionate+Formoterol fumarate+Glycopyrrolate bromide is effective for the treatment of severe COPD patients (chronic obstructive pulmonary disease)

DETAILED DESCRIPTION:
A 52-WEEK, DOUBLE BLIND, DOUBLE DUMMY, RANDOMIZED, 3-ARM PARALLEL GROUP, ACTIVE CONTROLLED CLINICAL TRIAL OF FIXED COMBINATION OF BECLOMETASONE DIPROPIONATE PLUS FORMOTEROL FUMARATE PLUS GLYCOPYRROLATE BROMIDE ADMINISTERED VIA PMDI (CHF 5993) VERSUS TIOTROPIUM BROMIDE AND VERSUS FIXED COMBINATION OF BECLOMETASONE DIPROPIONATE PLUS FORMOTEROL FUMARATE ADMINISTERED VIA PMDI AND TIOTROPIUM BROMIDE IN PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE

A total of 8 clinic visits (V0 to V7) will be performed during the study, as follows:

* A pre-screening visit (V0) to obtain the written informed consent from the patient
* A screening visit (V1) to establish the eligibility of patients, followed by a 2-week open-label run-in under Tiotropium
* After the randomisation (V2), patients will be assessed after 4, 12, 26, 40 and 52 weeks of treatment (V3 to V7) The assessments performed at visits include routine haematology and blood chemistry, medical history, physical examination, a 12-lead ECG, spirometric parameters, vital signs).

During the run-in and the randomised treatment periods, patients use an e-diary to record symptoms, rescue medication use and compliance to the study medications daily.

AEs/SAEs and COPD exacerbations will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male and female COPD patients aged ≥ 40 years
* Current smokers or ex-smokers
* FEV1<50% predicted (FEV1/FVC <0,7)
* at least 1 documented exacerbations in the last 12 Mo

Exclusion Criteria:

* Pregnant or lactating women and all women physiologically capable of becoming pregnant
* Diagnosis of asthma, history of allergic rhinitis or atopy
* Patients treated for exacerbations 1 Mo prior to screening
* Patients treated with non-cardioselective β-blockers
* Patients treated with long-acting antihistamines
* Known respiratory disorders other than COPD
* Patients who have clinically significant cardiovascular condition

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3686 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
COPD exacerbation rate | 52 weeks
  Moderate and severe COPD exacerbation rate over 52 weeks of treatment.

SECONDARY OUTCOMES:
pre-dose morning FEV1 | 52 weeks
  Change from baseline in pre-dose morning FEV1 at Week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen Vestbo, MD, Principal Investigator — Respiratory Research Group, Wythenshawe Hospital, MANCHESTER
Locations (3):
- Institut für klinische Forschung, Hessen, Germany
- Csongrád Megyei Mellkasi Betegségek Szakkórháza, Szeged, Hungary
- Azienda Ospedaliera Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Background] Vanfleteren L, Fabbri LM, Papi A, Petruzzelli S, Celli B. Triple therapy (ICS/LABA/LAMA) in COPD: time for a reappraisal. Int J Chron Obstruct Pulmon Dis. 2018 Dec 12;13:3971-3981. doi: 10.2147/COPD.S185975. eCollection 2018. PMID 30587953
- [Background] Singh D, Fabbri LM, Vezzoli S, Petruzzelli S, Papi A. Extrafine triple therapy delays COPD clinically important deterioration vs ICS/LABA, LAMA, or LABA/LAMA. Int J Chron Obstruct Pulmon Dis. 2019 Feb 28;14:531-546. doi: 10.2147/COPD.S196383. eCollection 2019. PMID 30880943
- [Background] Singh D, Fabbri LM, Corradi M, Georges G, Guasconi A, Vezzoli S, Petruzzelli S, Papi A. Extrafine triple therapy in patients with symptomatic COPD and history of one moderate exacerbation. Eur Respir J. 2019 May 18;53(5):1900235. doi: 10.1183/13993003.00235-2019. Print 2019 May. PMID 30792343
- [Result] Vestbo J, Papi A, Corradi M, Blazhko V, Montagna I, Francisco C, Cohuet G, Vezzoli S, Scuri M, Singh D. Single inhaler extrafine triple therapy versus long-acting muscarinic antagonist therapy for chronic obstructive pulmonary disease (TRINITY): a double-blind, parallel group, randomised controlled trial. Lancet. 2017 May 13;389(10082):1919-1929. doi: 10.1016/S0140-6736(17)30188-5. Epub 2017 Apr 3. PMID 28385353
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-000063-91/results
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-1208-PR-0090.pdf